CLINICAL TRIAL: NCT02107677
Title: Determination of Estimated Specificity of DENV Detect NS1 ELISAs
Brief Title: Specificity Study of Diagnostic for Early Detection of Dengue Infection
Status: Completed | Type: Observational
Sponsor: InBios International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DSC0094
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum

SUMMARY:
This study assesses the specificity of DENV Detect™ NS1 ELISA versus standard reference tests (e.g. PCR or viral culture) for dengue diagnosis in the US.

DENV Detect™ NS1 ELISA serves as an aid in the clinical laboratory diagnosis of early stages of Dengue infection in patients with clinical symptoms consistent with Dengue infection. This test is intended to be used on sera obtained within the first 7 days of symptoms. DENV Detect™ NS1 ELISA and rapid test results (positive or negative) must be confirmed by testing with a reference standard test.

This study will use archived, leftover human serum samples that have been sequentially collected from areas non-endemic for Dengue infection. Each specimen must have been collected within the first 7 days of symptoms, and must be accompanied by clinical data demonstrating that the individual had symptoms consistent with Dengue infection. The samples will have no personally identifiable information.

ELISAs and reference tests will be performed by different operators who are laboratory staff members. These staff members, blinded to each other's results, will evaluate the samples from each method independently.

ELIGIBILITY:
Inclusion Criteria:

* All age groups and both sexes.
* Serum samples collected within 1- 7 days of onset of symptoms consistent with Dengue virus infection.
* Information must be available about symptoms, age, and sex of patients from which samples are collected.

Exclusion Criteria:

* Any sample(s) with linked personal identifiers or any sample for which personal information can be discovered will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Human males and females of varying ages and geographical locations where dengue fever is non-endemic. We will use retrospective (archived) human serum samples, not collected specifically for this study and not individually identifiable to the Investigators. These samples will fall under the category of "leftover" specimens as described by FDA guidance. These archived samples will have been collected from patients within 7 days after onset of symptoms consistent with Dengue infection.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
number of subjects with negative result | one day

CONTACTS AND LOCATIONS:
Locations (1):
- State of Florida Dept. of Health Bureau of Laboratories Virology, Jacksonville, Florida, United States